CLINICAL TRIAL: NCT05264584
Title: Renoprotective Effect of Febuxostat on Contrast Induced Acute Kidney Injury in Chronic Kidney Disease Patients Stage 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MS 616/2020
Record Dates: First submitted 2022-02-18; First posted 2022-03-03 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-02

CONDITIONS: Chronic Kidney Disease stage3; Contrast-induced Nephropathy
MeSH Terms: interventions — Sodium Chloride; Acetylcysteine; Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control arm (Other): This arm is consisted of 60 patients.They will receive IV hydration and N-acetylcysteine (control arm).
  Interventions: Drug: Isotonic saline; Drug: N-acetyl cysteine
- Febuxostat arm (Experimental): This arm is consisted of 60 patients.They will receive IV hydration, N-acetylcysteine and Febuxostat .
  Interventions: Drug: Isotonic saline; Drug: N-acetyl cysteine; Drug: Febuxostat 80 MG

INTERVENTIONS:
Drug: Isotonic saline — All patients will receive a continuous intravenous infusion of isotonic saline at a rate of 0.5 mL/kg/h for at least 2 to 12 hours before the procedure and continued to receive it 6 to 24 hours afterward.
  Other Names: Saline
Drug: N-acetyl cysteine — all the patients will receive 600 mg orally twice daily ,on the day before and the day of exposure to contrast or a single periprocedural dose (within 4 hours of contrast exposure) 1200 mg .
  Other Names: NAC
Drug: Febuxostat 80 MG — All patients will receive a continuous intravenous infusion of isotonic saline at a rate of 0.5 mL/kg/h for at least 2 to 12 hours before the procedure and continued to receive it 6 to 24 hours afterward.
  Other Names: Feburic 80
  Arms: Febuxostat arm

SUMMARY:
This study will determine the renoprotective effect of febuxostat in prevention of contrast induced acute kidney injury in chronic kidney disease patients Stage 3 undergoing percutaneous coronary intervention.

DETAILED DESCRIPTION:
In this randomised non blinded clinical trial, Investigators will study 120 CKD patients undergoing PCI to determine the renoprotective effect of febuxostat in prevention of contrast induced acute kidney injury . So, the patients will be divided into two arms based on block randomization. Each arm compromise 60 patients. The first arm will receive IV hydration and N-acetylcysteine (ctrl arm) . The second arm will receive IV hydration, N-acetylcysteine and Febuxostat (F arm).

Block randomization will be used in this clinical trial design to reduce bias and achieve balance in the allocation of participants to treatment arms.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years old .

Patients under treatment of high dose statin(Atorvastatin (40-80 mg/day) .

Glomerular filtration rate=30-59ml/min.

Undergoing coronary PCI.

Exclusion Criteria:

Patients under treatment with febuxostat. Known allergy to febuxostat. High osmolar contrast media during the procedure .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
prevention of CI-AKI | 48-72 hours post contrast
  incidence of CI-AKI after 48-72 hours after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Rania Saad, Bachelor, Principal Investigator — Faculty of medicine Ain shams university; Iman Sarhan, PhD, Study Director — Faculty of medicine Ain Shams university; Nahla Teama, PhD, Study Chair — Faculty of medicine Ain Shams university; Yasser Alaa, PhD, Study Chair — Faculty of medicine Ain Shams university
Locations (1):
- Ain shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol